CLINICAL TRIAL: NCT00160693
Title: A Phase III, Multicenter, Open-Label Long-Term Study to Assess the Safety and Tolerability of CDP870 400 mg Subcutaneously Every 4 Weeks, in Subjects With Rheumatoid Arthritis
Brief Title: Open Label Long-Term Safety Study of Certolizumab Pegol (CZP) for Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C87015; 2005-002617-21 (EudraCT Number)
Expanded Access: NCT03559686 (Available)
Record Dates: First submitted 2005-09-06; First posted 2005-09-12 (Estimated); Results first posted 2012-07-09 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; America College of Rheumatology; Disease modifying anti-rheumatic drug; Certolizumab Pegol (CDP870)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Certolizumab Pegol (Experimental)
  Interventions: Biological: Certolizumab Pegol

INTERVENTIONS:
Biological: Certolizumab Pegol — 400 mg of Certolizumab Pegol subcutaneously every 4 Weeks
  Other Names: Cimzia

SUMMARY:
The primary purpose of this study is to obtain long-term safety data with CZP in patients with Rheumatoid Arthritis (RA). Additional objectives are to assess the dose and type of Arthritis medication(s) utilized by patients, and to assess the long-term impact of CZP on physical function. Treatment will continue up to approval of a marketing application for this product.

ELIGIBILITY:
Inclusion Criteria:

* Participation in CZP trial C87014 or C87011
* If female and of childbearing potential, she agrees to participate in this study by providing written informed consent, has been using adequate contraception since her last menses, will use adequate contraception during the study and for 12 weeks after the last dose of study drug (or longer if required by local regulations), is not lactating, and has had a negative urine pregnancy test on the day of receiving the first dose of study drug
* Must have provided written informed consent before undergoing any study procedures

Exclusion Criteria:

* History (Hx) of chronic infection, serious or life-threatening infection - (including Herpes Zoster) within 6 months prior, or any current symptom indicating infection
* Current or recent Hx of severe, progressive and/or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological or cerebral disease
* Any finding indicative of Tuberculosis at end of previous study
* Known HIV infection
* Persistently abnormal AST (Aspartate Aminotransferase) or ALT (Alanine Aminotransferase) results (> 2 times upper limit of normal)
* Hemoglobin (Hgb) levels < 9 g/dL or Hematocrit < 30 %
* Total White Blood Cell (WBC) count of < 3.0 x 100/L (< 3000/mm^3)
* Platelet count < 100 x 100 L (100,000/mm^3)
* Serum creatinine > 1.5 times upper limit of normal based on patient age and sex
* Receipt of any biological therapies for RA in 6 months prior to study entry or any prior treatment (tx) with Tumor Necrosis Factor (TNF) blocking agent (excluding CDP870)
* Receipt of any vaccination (live, attenuated or killed) in 8 weeks prior to Baseline
* Any other condition which the Principal Investigator judges would make patient unsuitable for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2003-03; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (61):
- United States (29):
  - Huntsville, Alabama
  - Paradise Valley, Arizona
  - Washington D.C., District of Columbia
  - Aventura, Florida
  - Clearwater, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Coeur d'Alene, Idaho
  - Springfield, Illinois
  - Wichita, Kansas
  - Wheaton, Maryland
  - Fall River, Massachusetts
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Charlotte, North Carolina
  - Cleveland, Ohio
  - Dayton, Ohio
  - Erie, Pennsylvania
  - West Reading, Pennsylvania
  - Charleston, South Carolina
  - Memphis, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Duncanville, Texas
  - Lubbock, Texas
  - San Antonio, Texas
  - San Diego, Texas
  - Everett, Washington
- Austria (3):
  - Graz
  - Klagenfurt
  - Vienna
- Belgium (4):
  - Antwerp
  - Diepenbeek
  - Liège
  - Merksem
- Czechia (6):
  - České Budějovice
  - Liberec
  - Ostrava Trebovice
  - Prague
  - Praha4 -KRC
  - Uherské Hradiště
- Germany (7):
  - Berlin
  - Cologne
  - Gortlitz
  - Hamburg
  - Jena
  - Leipzig
  - Ratingen
- Ireland (2):
  - Dublin
  - Waterford
- United Kingdom (10):
  - Birmingham
  - Cannock
  - Colchester
  - Glasgow
  - Harrogate
  - London
  - Manchester
  - Metropolitan Borough of Wirral
  - Oxford
  - Peterborough

REFERENCES:
- [Result] Fleischmann R, van Vollenhoven RF, Vencovsky J, Alten R, Davies O, Mountian I, de Longueville M, Carter D, Choy E. Long-Term Maintenance of Certolizumab Pegol Safety and Efficacy, in Combination with Methotrexate and as Monotherapy, in Rheumatoid Arthritis Patients. Rheumatol Ther. 2017 Jun;4(1):57-69. doi: 10.1007/s40744-017-0060-8. Epub 2017 Mar 28. PMID 28353191
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects must have participated in CZP trial C87011 [NCT00548834] or C87014 [NCT00544154] for at least 12 weeks to be eligible to enter the study.
  All enrolled subjects who received at least one dose of study medication are included in the Safety Set (SS).
Pre-assignment Details: Participant Flow and Baseline Characteristics refer to the Safety Set (SS). Baseline Characteristics were measured at Baseline of the respective feeder study.
Period: Overall Study
Arm/Group | Certolizumab Pegol
Started | 402
Completed | 167
Not Completed | 235
Not completed — Adverse Event | 97
Not completed — Lack of Efficacy | 30
Not completed — Protocol Violation | 24
Not completed — Lost to Follow-up | 15
Not completed — Withdrawal by Subject | 54
Not completed — Study terminated by sponsor | 15

BASELINE CHARACTERISTICS:
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 402
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 327
  >=65 years | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 303
  Male | 99
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 363
  More than one race | 0
  Unknown or Not Reported | 17
Region of Enrollment [Number; unit: participants]
  United States | 160
  Czech Republic | 81
  Belgium | 11
  Ireland | 8
  Austria | 19
  Germany | 87
  United Kingdom | 36
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 78.00 (17.88)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 166.4 (8.6)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram/ meter^2 (kg / m^2)] — The BMI was calculated as: Weight (kg)/(Height(cm)/100)^2
  kilogram/ meter^2 (kg / m^2) | 28.20 (6.34)
Disease Duration [Mean (Standard Deviation); unit: years] | 9.46 (8.13)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With at Least One Adverse Event (AE) During the Study Period of 8 Years
Description: An AE is any untoward medical occurrence in a subject or trial subject that is administered a drug or biologic (medicinal product) or that is using a medical device. The event does not necessarily have a causal relationship with that treatment or usage.
  First dose of CZP was at Baseline of one of the feeder studies C87011 [NCT00548834] or C87014 [NCT00544154] for subjects randomized to CZP, or at First Visit (Week 0) of this study for subjects randomized to Placebo.
Time Frame: From first dose of CZP up to 8 years
Population: Safety Set (SS).
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 402
percentage of subjects | 93.5

2. Primary Outcome: Percentage of Subjects Who Withdrew Due to an Adverse Event (AE) During the Study Period of 8 Years
Description: An AE is any untoward medical occurrence in a subject or trial subject that is administered a drug or biologic (medicinal product) or that is using a medical device. The event does not necessarily have a causal relationship with that treatment or usage.
  The results of this Primary Outcome Measure are summarized from the Adverse Event pages of the Case Report Forms.
Time Frame: From First Visit (Week 0 in this study) up to 8 years
Population: Safety Set (SS).
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 402
percentage of subjects | 24.9

3. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 20% Response Criteria (ACR20) at Week 52
Description: The assessments are based on a 20% or greater improvement from Baseline to Week 52 in the number of tender joints, a 20% or more improvement in the number of swollen joints, and a 20% or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP).
  Baseline is Baseline of the respective feeder study.
Time Frame: From Baseline to Week 52
Population: Of the 402 subjects in the Safety Set (SS), 370 subjects are included in this analysis, because they had available data at Baseline and Week 52.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 370
percentage of subjects | 58.1 [53.1 to 63.1]

4. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 20% Response Criteria (ACR20) at Week 100
Description: The assessments are based on a 20% or greater improvement from Baseline to Week 100 in the number of tender joints, a 20% or more improvement in the number of swollen joints, and a 20% or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP).
  Baseline is Baseline of the respective feeder study.
Time Frame: From Baseline to Week 100
Population: Of the 402 subjects in the Safety Set (SS), 275 subjects are included in this analysis, because they had available data at Baseline and Week 100.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 275
percentage of subjects | 60.0 [54.2 to 65.8]

5. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 20% Response Criteria (ACR20) at Week 160
Description: The assessments are based on a 20% or greater improvement from Baseline to Week 160 in the number of tender joints, a 20% or more improvement in the number of swollen joints, and a 20% or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP).
  Baseline is Baseline of the respective feeder study.
Time Frame: From Baseline to Week 160
Population: Of the 402 subjects in the Safety Set (SS), 247 subjects are included in this analysis, because they had available data at Baseline and Week 160.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 247
percentage of subjects | 68.4 [62.6 to 74.2]

6. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 20% Response Criteria (ACR20) at Week 208
Description: The assessments are based on a 20% or greater improvement from Baseline to Week 208 in the number of tender joints, a 20% or more improvement in the number of swollen joints, and a 20% or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP).
  Baseline is Baseline of the respective feeder study.
Time Frame: From Baseline to Week 208
Population: Of the 402 subjects in the Safety Set (SS), 223 subjects are included in this analysis, because they had available data at Baseline and Week 208.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 223
percentage of subjects | 72.6 [66.8 to 78.5]

7. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 20% Response Criteria (ACR20) at Week 256
Description: The assessments are based on a 20% or greater improvement from Baseline to Week 256 in the number of tender joints, a 20% or more improvement in the number of swollen joints, and a 20% or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP).
  Baseline is Baseline of the respective feeder study.
Time Frame: From Baseline to Week 256
Population: Of the 402 subjects in the Safety Set (SS), 211 subjects are included in this analysis, because they had available data at Baseline and Week 256.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 211
percentage of subjects | 75.4 [69.5 to 81.2]

8. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 20% Response Criteria (ACR20) at Week 316
Description: The assessments are based on a 20% or greater improvement from Baseline to Week 316 in the number of tender joints, a 20% or more improvement in the number of swollen joints, and a 20% or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP).
  Baseline is Baseline of the respective feeder study.
Time Frame: From Baseline to Week 316
Population: Of the 402 subjects in the Safety Set (SS), 140 subjects are included in this analysis, because they had available data at Baseline and Week 316.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 140
percentage of subjects | 76.4 [69.4 to 83.5]

9. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 20% Response Criteria (ACR20) at Completion Visit or Early Withdrawal Visit
Description: The assessments are based on a 20% or greater improvement from Baseline to the Completion Visit or early Withdrawal Visit in the number of tender joints, a 20% or more improvement in the number of swollen joints, and a 20% or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP).
Time Frame: From Baseline to Completion Visit/ early Withdrawal Visit, up to 8 years
Population: Safety Set (SS).
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 402
percentage of subjects | 57.2 [52.4 to 62.1]

10. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 50% Response Criteria (ACR50) at Completion Visit or Early Withdrawal Visit
Description: The assessments are based on a 50% or greater improvement from Baseline to the Completion Visit or early Withdrawal Visit in the number of tender joints, a 50% or more improvement in the number of swollen joints, and a 50% or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP).
Time Frame: From Baseline to Completion Visit/ early Withdrawal Visit, up to 8 years
Population: Safety Set (SS).
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 402
percentage of subjects | 27.6 [23.2 to 32.0]

11. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 70% Response Criteria (ACR70) at Completion Visit or Early Withdrawal Visit
Description: The assessments are based on a 70% or greater improvement from Baseline to the Completion Visit or early Withdrawal Visit in the number of tender joints, a 70% or more improvement in the number of swollen joints, and a 70% or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP).
Time Frame: From Baseline to Completion Visit/ early Withdrawal Visit, up to 8 years
Population: Safety Set (SS).
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 402
percentage of subjects | 7.7 [5.1 to 10.3]

12. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ- DI) at Completion Visit or Early Withdrawal Visit
Description: The HAQ-DI assesses the degree of difficulty experienced in eight domains (Dressing and Grooming, Arising, Eating, Walking, Hygiene, Reach, Gripping, Other Activities) of daily living activities using 20 questions. The HAQ-DI is calculated by summing the domain scores and dividing them by the number of domains. It ranges from 0 (no difficulty) to 3 (unable to do). Negative values indicate an improvement from Baseline to the Post-Baseline Visit with larger negative values showing a better improvement.
Time Frame: From Baseline to Completion Visit/ early Withdrawal Visit, up to 8 years
Population: Of the 402 subjects in the Safety Set (SS), 400 subjects are included in this analysis, because they had available data at Baseline and Completion or early Withdrawal Visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 400
units on a scale | -0.305 (0.620)

13. Secondary Outcome: Percentage of Subjects Who Withdrew Due to Lack of Efficacy During the Study Period of 8 Years
Time Frame: From First Visit (Week 0 in this study) up to 8 years
Population: Safety Set (SS).
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 402
percentage of subjects | 7.5

14. Secondary Outcome: Percentage of Subjects Utilizing Common Additional Arthritis Medications During the Study Period of 8 Years
Description: This Secondary Outcome Measure shows additional arthritis medications received by at least 20% of subjects during the 8-year study.
Time Frame: From First Visit (Week 0 in this study) up to 8 years
Population: Safety Set (SS).
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 402
percentage of subjects
  Acetylsalicylic acid | 21.9
  Celecoxib | 22.9
  Diclofenac | 23.4
  Folic acid | 65.2
  Ibuprofen | 26.4
  Methotrexate | 60.9
  Methylprednisolone | 33.8
  Other Immunosuppressive agents | 25.9
  Paracetamol | 29.6
  Prednisolone | 20.4
  Prednisone | 39.3

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected over the whole Study Period of 8 Years from first dose of study medication (Baseline of feeder study or First Visit of this study for subjects randomized to Placebo) to 24 Weeks post last dose (Last Follow-up Visit).
Description: AEs refer to the Safety Set (SS). SS includes all of the 402 enrolled subjects.
Arm/Group | Certolizumab Pegol
Serious Adverse Events (participants affected / at risk) | 184/402
Other Adverse Events (participants affected / at risk) | 348/402
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (N=402)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 2 (2)
Abscess intestinal (Infections and infestations) | 1 (1)
Abscess neck (Infections and infestations) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2)
Acute prerenal failure (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (3)
Angina pectoris (Cardiac disorders) | 3 (3)
Angina unstable (Cardiac disorders) | 2 (2)
Aortic aneurysm (Vascular disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (2)
Arterial occlusive disease (Vascular disorders) | 1 (1)
Arterial stenosis (Vascular disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthritis infective (Infections and infestations) | 1 (1)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 4 (5)
Atrioventricular block (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2)
Bile duct stone (Hepatobiliary disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Bronchitis (Infections and infestations) | 3 (3)
Bronchitis acute (Infections and infestations) | 1 (1)
Bronchopneumonia (Infections and infestations) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 4 (4)
Cellulitis (Infections and infestations) | 4 (9)
Cerebral ischaemia (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 3 (6)
Chest pain (General disorders) | 3 (4)
Chills (General disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 2 (2)
Cholangitis suppurative (Infections and infestations) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 3 (3)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 3 (3)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Chronic sinusitis (Infections and infestations) | 1 (1)
Chronic tonsillitis (Infections and infestations) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1)
Clostridial infection (Infections and infestations) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Contrast media reaction (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Coronary artery disease (Cardiac disorders) | 6 (6)
Coronary artery stenosis (Cardiac disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Device failure (Injury, poisoning and procedural complications) | 1 (2)
Device related infection (Infections and infestations) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1)
Diverticulum duodenal (Gastrointestinal disorders) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Empyema (Infections and infestations) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2)
Escherichia sepsis (Infections and infestations) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (4)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Finger deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 2 (2)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1)
Foreign body trauma (Injury, poisoning and procedural complications) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastritis erosive (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3)
Gastroenteritis clostridial (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Global amnesia (Nervous system disorders) | 1 (1)
Goitre (Endocrine disorders) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hepatitis cholestatic (Hepatobiliary disorders) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 2 (2)
Hilar lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Histoplasmosis disseminated (Infections and infestations) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Hypertensive crisis (Vascular disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1)
Impaired healing (General disorders) | 2 (4)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1)
Incontinence (Renal and urinary disorders) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Inflammatory bowel disease (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 2 (2)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 (4)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Joint destruction (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Leukoplakia oral (Gastrointestinal disorders) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lymph node tuberculosis (Infections and infestations) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 2 (2)
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Maculopathy (Eye disorders) | 1 (1)
Malaise (General disorders) | 1 (2)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mastitis (Infections and infestations) | 1 (1)
Medical device complication (Injury, poisoning and procedural complications) | 1 (1)
Medication error (Injury, poisoning and procedural complications) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1)
Mixed incontinence (Renal and urinary disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 5 (5)
Myocardial ischaemia (Cardiac disorders) | 2 (2)
Necrotising fasciitis (Infections and infestations) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 4 (5)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Oedematous pancreatitis (Gastrointestinal disorders) | 1 (1)
Oesophageal rupture (Gastrointestinal disorders) | 1 (1)
Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Optic nerve disorder (Eye disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 16 (21)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Panic disorder (Psychiatric disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1)
Pelvic abscess (Infections and infestations) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Perforation bile duct (Hepatobiliary disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 9 (10)
Pneumonia legionella (Infections and infestations) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pubic rami fracture (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pulmonary tuberculosis (Infections and infestations) | 1 (1)
Purulent synovitis (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Pyrexia (General disorders) | 3 (3)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Rectocele (Reproductive system and breast disorders) | 1 (1)
Renal cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 16 (20)
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Stress incontinence (Renal and urinary disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 2 (3)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (3)
Synovectomy (Surgical and medical procedures) | 1 (2)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovial rupture (Injury, poisoning and procedural complications) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 2 (3)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
Thyroid gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Toe deformity (Musculoskeletal and connective tissue disorders) | 5 (5)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tonsillitis (Infections and infestations) | 2 (2)
Tracheobronchitis (Infections and infestations) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
XIth nerve injury (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (N=402)
Abdominal pain upper (Gastrointestinal disorders) | 22 (31)
Alanine aminotransferase increased (Investigations) | 27 (34)
Anaemia (Blood and lymphatic system disorders) | 25 (31)
Arthralgia (Musculoskeletal and connective tissue disorders) | 65 (118)
Back pain (Musculoskeletal and connective tissue disorders) | 90 (137)
Bronchitis (Infections and infestations) | 58 (89)
Bronchitis acute (Infections and infestations) | 25 (45)
Bursitis (Musculoskeletal and connective tissue disorders) | 28 (40)
Conjunctivitis (Eye disorders) | 29 (34)
Constipation (Gastrointestinal disorders) | 24 (29)
Contusion (Injury, poisoning and procedural complications) | 30 (44)
Cough (Respiratory, thoracic and mediastinal disorders) | 82 (126)
Cystitis (Infections and infestations) | 33 (45)
Depression (Psychiatric disorders) | 39 (49)
Diarrhoea (Gastrointestinal disorders) | 64 (135)
Dizziness (Nervous system disorders) | 42 (59)
Dyspepsia (Gastrointestinal disorders) | 41 (60)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 (32)
Fall (Injury, poisoning and procedural complications) | 28 (42)
Fatigue (General disorders) | 65 (86)
Headache (Nervous system disorders) | 86 (135)
Herpes simplex (Infections and infestations) | 44 (70)
Herpes zoster (Infections and infestations) | 24 (27)
Hypertension (Vascular disorders) | 78 (94)
Influenza (Infections and infestations) | 40 (56)
Insomnia (Psychiatric disorders) | 36 (44)
Joint swelling (Musculoskeletal and connective tissue disorders) | 21 (39)
Lower respiratory tract infection (Infections and infestations) | 27 (65)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 27 (34)
Nasopharyngitis (Infections and infestations) | 141 (380)
Nausea (Gastrointestinal disorders) | 49 (65)
Neck pain (Musculoskeletal and connective tissue disorders) | 22 (26)
Oedema peripheral (General disorders) | 38 (54)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 26 (49)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 46 (68)
Paraesthesia (Nervous system disorders) | 23 (29)
Pharyngitis (Infections and infestations) | 21 (36)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 38 (52)
Rash (Skin and subcutaneous tissue disorders) | 66 (104)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 63 (109)
Sciatica (Nervous system disorders) | 28 (34)
Sinusitis (Infections and infestations) | 74 (123)
Upper respiratory tract infection (Infections and infestations) | 93 (198)
Urinary tract infection (Infections and infestations) | 84 (159)
Viral infection (Infections and infestations) | 27 (42)
Vomiting (Gastrointestinal disorders) | 37 (58)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days